CLINICAL TRIAL: NCT06967337
Title: Short, Animated Storytelling Video and Written Messages to Promote Adoption of Health "Microsteps": an Online Randomized Experiment
Brief Title: Microsteps Study-Short, Animated Storytelling Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Maya Adam, Clinical Associate Professor in Department of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 80047
Record Dates: First submitted 2025-05-02; First posted 2025-05-13 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Behavior, Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Written messages of Microsteps and Instructional video (Experimental): Participants will be shown written Microsteps messages presenting various behavioral nudges and a short instructional video. Thereafter, they will be asked to complete a questionnaire to assess their behavioral expectation of adopting the behavioral nudges and two visual analogue scales measuring hope and happiness. Two weeks later, participants will be invited to return and complete these outcome assessments again.
  Interventions: Behavioral: Microsteps; Behavioral: Instructional Video
- Written messages of Microsteps and Storytelling video (Experimental): Participants will be shown written Microsteps messages presenting various behavioral nudges, as well as a short, animated storytelling video. Thereafter, they will be asked to complete the questionnaire assessing their behavioral expectation of adopting the behavioral nudges and two visual analogue scales measuring hope and happiness. Two weeks later, participants will be invited to return and complete these outcome assessments again.
  Interventions: Behavioral: Microsteps; Behavioral: Storytelling video
- Do-nothing Control Group (No Intervention): Participants will not be exposed to either the microsteps or video content before they are asked to complete the questionnaire assessing their behavioral expectation of adopting the behavioral nudges and two visual analogue scales measuring hope and happiness. Two weeks later, participants will be invited to return and complete these outcome assessments again.

INTERVENTIONS:
Behavioral: Microsteps — Microsteps (behavioral nudges) are a series of short, written messages that were developed by the Thrive Global Wellbeing and Behavior Change Platform, based in the US. The Microsteps messages deliver step-wise, small health behavioral nudges that align with research on behavior change strategies. The behavioral nudges focus on health behaviors that could be useful adjunct interventions for GLP-1RA users, (improved food choices, exercise, sleep and stress management).
  Arms: Written messages of Microsteps and Instructional video; Written messages of Microsteps and Storytelling video
Behavioral: Storytelling video — The storytelling video is a short, 2D animated, wordless storytelling video, of 2:21 minutes duration. The humorous, animated story features a minion-like character who, with the help of their dog, learns to adopt better health behaviors after experiencing an episode of burnout. The video mirrors the written Microsteps messages, conveying them through comical demonstration, rather than through instructional language. The animated characters are free of cultural identifiers, with the intention of increasing the accessibility of the video by overcoming barriers associated with culture, education, language and literacy. The video is intended to underscore and complement the written Microsteps messages, enhance their durability and boost hope and happiness in viewers.
  Arms: Written messages of Microsteps and Storytelling video
Behavioral: Instructional Video — The Instructional Video is a short 2:27min video demonstrating the microsteps and presenting additional information about the rationale for adopting them. The video features an educator who explains these points in a didactic format, and a second educator who demonstrates performing a microstep (stretching at a desk).
  Arms: Written messages of Microsteps and Instructional video

SUMMARY:
This study evaluates the effect of single exposure to written Microsteps messages and short video booster content, on behavioral expectation to adopt behavioral nudges, in the immediate and medium term. Beyond that, the study will examine the effect of exposure to written Microsteps messages and short video booster content, on hope and happiness. This study will be conducted entirely online. Adult participants, in the US and the UK, will be recruited through the platform Prolific Academic (ProA).

ELIGIBILITY:
Inclusion Criteria:

* Registered with the Prolific Academic platform
* Using a GLP-1RA medication or having used a GLP-1RA medication in the past.

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5431 (Actual)
Dates: Start 2025-06-19 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Effects of the written Microsteps, with instructional booster video or storytelling booster video, on behavioral expectation to adopt behavioral nudges, in the immediate and medium-term. | Baseline, immediately post-intervention exposure (up to 24 hours) and 2 weeks post exposure.
  This measure is intended to explore the effect of the written messages, with two different approaches to the video booster, on behavioral expectation to adopt the Microsteps, in the immediate and medium-term. The Microsteps questionnaire consists of 8 questions, each measured on a Likert scale from 1-5 where 1 = very unlikely and 5 = very likely.

SECONDARY OUTCOMES:
Medium-term effects of the written Microsteps, with instructional booster video or storytelling booster video, on self-reported consumption of sweetened beverages. | Baseline, 2 weeks post intervention exposure
  Participants self report frequency of consuming sugar-sweetened drinks at baseline and two weeks after single exposure to the written Microsteps, with instructional booster video or storytelling booster video. Participants are asked how often they choose to drink sugar-sweetened drinks on a 4-item scale from never/rarely to daily.
Medium-term effects of the written Microsteps, with instructional booster video or storytelling booster video, on self-reported consumption of dietary protein. | Baseline, 2 weeks post intervention exposure
  Participants self report frequency of including protein-rich foods in each of their meals, at baseline and two weeks after single exposure to the written Microsteps, with instructional booster video or storytelling booster video. Participants are asked how often they include protein-rich foods in each of their meals, on a 4-item scale from never/rarely to daily.
Medium-term effects of the written Microsteps, with instructional booster video or storytelling booster video, on self-reported physical activity. | Baseline, 2 weeks post intervention exposure
  Participants self report frequency of including protein-rich foods in each of their meals, at baseline and two weeks after single exposure to the written Microsteps, with instructional booster video or storytelling booster video. Participants are asked how often they engage in physical activity that gets their heart rate up, on a 4-item scale from never/rarely to daily.
Effects of the written Microsteps, with instructional booster video or storytelling booster video, on Hope | Baseline, immediately post intervention exposure (up to 24 hours) and 2 weeks post intervention exposure
  Participants self-report levels of hope using a visual analogue scale (VAS), a longstanding, validated tool for assessing related constructs of stress and subjective well-being.The scale goes from zero to 100 and higher scores indicate higher levels of hope.
Effects of the written Microsteps, with instructional booster video or storytelling booster video, on Happiness | Baseline, immediately post intervention exposure (up to 24 hours) and 2 weeks post intervention exposure
  Participants self-report levels of happiness on VAS, a longstanding, validated tool for assessing related constructs of stress and subjective well-being

CONTACTS AND LOCATIONS:
Overall Officials: Maya Adam, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No